CLINICAL TRIAL: NCT00578149
Title: Bevacizumab and Carboplatin/Paclitaxel and Radiation in Stage III Non-Small Cell Lung Cancer
Brief Title: Bevacizumab and Carboplatin/Paclitaxel and Radiation in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-415
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: chemoradiotherapy; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Bevacizumab; Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
This study is being done to learn what effects (good and bad) bevacizumab in conjunction with carboplatin/paclitaxel and radiation therapy has on patients with non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
* There are three phases of treatment 1)chemoradiation, 2) consolidation and 3)maintenance therapy.
* The chemoradiation phase is from week 1 to week 7. The following will occur during this phase: Daily chest radiation starting on day 1; pre-medication for paclitaxel; weekly intravenous administration of paclitaxel and carboplatin; intravenous administration of bevacizumab once weekly every three weeks starting on day 1.
* During weeks 8-9, patients will undergo a PET/CT scan for restaging.
* The consolidation phase is from week 10 to week 16. The following will occur during this phase: Pre-medication for paclitaxel; intravenous administration of paclitaxel and carboplatin twice weekly every 3 weeks; intravenous administration of bevacizumab once weekly every 3 weeks.
* The maintenance phase is from week 17 to week 52. The following will occur during this phase; intravenous administration of bevacizumab once a week every three weeks for 1 year; PET/CT scan every three months.
* The following evaluations will occur during treatment: 1)Patients will be evaluated weekly by the study doctor, 2) Weight, difficulty or discomfort in swallowing, shortness of breath and over well-being will be recorded, 3) Weekly lab test will include CBC, chemistries, and liver function tests. 4) Followed through each cycle of chemotherapy and every 6-8 weeks for the duration of the study.
* The following evaluations will occur after treatment: 1)Every 6-8 weeks assessed for response with a CT or PET/CT scan for one year, 2) Toxicity will also be assessed at each follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC) that have been evaluated and determined not to be candidates for surgical resection as part of their definitive management of stage III disease.
* Age 18 years or older
* ECOG performance status of 0-1
* Life Expectancy of greater than six months
* Normal organ and marrow function
* Women and men of child-bearing potential must agree to use adequate contraception

Exclusion Criteria:

* Prior chemotherapy or thoracic radiation therapy
* Squamous histology or any histology in close proximity to a major vessel
* Active hemoptysis
* History of hypercoagulability
* Known distant metastatic disease
* History of allergic reactions attributed to compounds with similar chemical or biological composition to bevacizumab, carboplatin, paclitaxel or other agents used in this study
* Patients with uncontrolled intercurrent illness
* Pregnant women
* Major surgical procedure, open biopsy, or significant traumatic injury with in 28 days prior to day 0
* Minor surgical procedure within 7 days to day 0
* HIV-positive patients receiving combination anti-retroviral therapy.
* Non-skin cancer malignancy in the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To examine the time to progression of the novel regimen in stage III patients treated with concurrent chemoradiotherapy.

SECONDARY OUTCOMES:
Response rate, overall survival, and patterns of failure and toxicity of the novel therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Allen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts